CLINICAL TRIAL: NCT04176978
Title: Effects of Tight-control Strategy With and Without Rosuvastatin on Progression of Subclinical Carotid and Coronary Atherosclerosis in Psoriatic Arthritis- a Randomized Controlled Study
Brief Title: PsA T2T Statin Trial on Carotid and Coronary Atherosclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2019.063T
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Psoriatic Arthritis; Atherosclerosis
MeSH Terms: conditions — Arthritis, Psoriatic; Atherosclerosis | interventions — Rosuvastatin Calcium; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T2T + statin (Experimental): Patient in this arm will receive treat-to-target strategy with rousavastin 20mg
  Interventions: Drug: Rosuvastatin; Other: Treat-to-target strategy
- T2T only (Active Comparator): Patient in this arm will receive treat-to-target strategy only.
  Interventions: Other: Treat-to-target strategy

INTERVENTIONS:
Drug: Rosuvastatin — Patient in this group will receive Rosuvastatin 20mg daily.
  Other Names: Statin
  Arms: T2T + statin
Other: Treat-to-target strategy — Patient will receive treat-to-target strategy aiming at minimal disease activity (MDA). If patient cannot achieve MDA, treatment will be escalated.
  Other Names: T2T

SUMMARY:
Psoriatic arthritis (PsA) is a chronic inflammatory disease associated with an increased risk of myocardial infarction (MI). Using coronary computer tomography angiogram (CCTA), it is found that a significantly higher prevalence of high-risk coronary plaque (non-calcified plaque [NCP]), supporting the notion that more aggressive cardiovascular (CV) evaluation strategy should be considered in these patients.

Carotid ultrasound screening in this population may be a better alternative than traditional risk score to identify patients at high CV risk as the latter underestimated CV risk. Previous study from our group have demonstrated that achieving treatment target (minimal disease activity [MDA]) can prevent progression of carotid atherosclerosis. Nevertheless, 38% of this Treat to Target (T2T) cohort still had carotid plaque progression.

Project description

it is hypothesized that combination of a T2T stratgy together with high-intensity rosuvastatin treatment (Group 1: T2T-statin group) is more effective in preventing progression of coronary and carotid atherosclerosis than T2T stratgy alone (Group 2: T2T-only group) in high-risk PsA patients with carotid plaque.

The primary outcome is to ascertain the effect of T2T strategy with high-intensity rosuvastain (Group 1: T2T-statin group) on the change in CIMT over a period of 12 months compared with T2T strategy alone (Group 2: T2T-only group)

DETAILED DESCRIPTION:
Treatment protocol This is a 1-year prospective, hospital-based, open-label, randomized, controlled trial. The trial comprised two arms. Group 1 will receive T2T strategy together with rosuvastain 20mg daily (T2T-statin group). Group 2 will receive T2T strategy only (T2T-only group). The method of concealed random allocation will be used. Simple randomization will be conducted by a computer-generated random list.

Use of statins The patients will be given the necessary number of rosuvastatin tablets at each visit. At the following visits, surplus medication will be returned to the investigator. Compliance is calculated as a percentage, based on the number of tablets returned.

No trials to date that have evaluated effects on CVD events have tested any medication in combination with statins or treatment to specific LDL-C goals, therefore we do not intensify the regimen for any particular level of LDL-C response. Measuring LDL-C response after initiating therapy in this study is mainly to assess adherence. In this primary prevention trial, in patients who do not tolerate statins, no lipid-lowering therapy will be administered. Potential interventions include lifestyle modification.

Use of DMARDs All participants will receive a 1-year protocolized treatment with the aim to achieve MDA. A predefined treatment protocol is developed based on the EULAR recommendations and the Hong Kong guideline for the use of bDMARDs. Patients fulfilling the criteria for bDMARDs can either pay out of pocket or can apply for the Samaritan Fund for financial assistance, provided they must pass a household-based financial assessment (http://www.ha.org.hk/visitor/ha_visitor_index.asp?content_id=212020). When patient cannot achieve treatment goal within 3-6 months of therapy, the treatment therapy will be escalated to the next step according to the protocol, unless the patient declined or toxic effects preclude this approach. For the introduction of DMARD only joint involvement is taken into account. The participants with active disease who failed non-steroidal anti-inflammatory drug (NSAID) or those with poor prognostic factor will start with methotrexate monotherapy, which is increased to 20mg/week or maximum tolerated dose. Subsequent steps for patients who fail to achieve treatment goal include switching to other conventional synthetic DMARDs (csDMARDs), combination csDMARD therapy or TNFi, ustekinumab, secukinumab or tofacitinib. Intra-articular steroid or local steroid injection to enthesitis and dactylitis are allowed during the study but will be forbidden in the 4 weeks before assessment.

Clinical Assessment Assessment performed at each visit include pain, physicians' and patients' global assessments, number of tender joints count (TJC) and swollen joints count (SJC) (using the 68 tender/66 SJC), Maastricht Ankylosing Spondylitis Enthesitis Score (MASES), number of digits with dactylitis; ankylosing spondylitis disease activity score (ASDAS), modified health assessment questionnaire (M-HAQ); Disease Activity index for Psoriatic Arthritis (DAPSA), Psoriasis Area (BSA), Psoriasis Activity and Severity Index (PASI) were used to measure joint and skin disease activity.(31) MDA was used for assessment of treatment efficacy endpoint. The MDA criteria assess 7 domains [TJC ≤ 1, SJC ≤ 1, enthesitis count ≤ 1, skin (≤ 1 or BSA ≤ 3%), function (measured by the Health Assessment Questionnaire), ≤ 0.5, patient's global VAS on a 100-mm scale ≤ 20, and patient pain VAS on a 100 mm scale ≤ 15]. If 5 of 7 of the cutoffs for these domains are met, then the patient is deemed to be in MDA.

Cardiovascular assessments The following anthropomorphic assessment will be performed at each visit. Anthropomorphic measurements include body heights, body weight, waist and hip circumferences, two consecutive blood pressure readings in sitting position and heart rate. Hypertension status is defined as systolic blood pressure (SBP) ≥140mmHg or diastolic blood pressure (DBP) ≥90mmHg or the use of antihypertensive agents. Other data include menopausal status, smoking and drinking habits, history of DM, hypertension, hypercholesterolemia, overt CVD, and family history of CVD, DM in first-degree male relatives <55 years of age or first-degree female relatives <65 years of age. Drug history is retrieved from case notes or elicited during the clinical assessment.

Laboratory assessments and inflammatory markers Laboratory assessments at each visit include complete blood count, liver and renal function tests, creatine kinase (CK), ESR and C-reactive protein (CRP), fasting blood glucose, lipid profile (total cholesterol [TC], LDL-C, high-density lipoprotein-cholesterol [HDL-C], triglycerides), fibrinogen and uric acid.

Carotid intima-media thickness (CIMT) and plaque CIMT and plaque will be assessed at baseline and 12 months.CIMT will be measured using a high-resolution B-mode ultrasound machine (Philips EPIQ7) by an experienced sonographer blinded to all clinical information using a 30-MHz linear vascular probe (Philips L12-3 broadband linear array transducer). The CIMT will be measured offline in the distal common carotid artery, bulb, and proximal internal carotid artery using dedicated software (Philips Xcelera Cardiology Enterprise Viewer Client 4). The mean and maximal IMT values of 6 arterial segments will be calculated for further analysis. Plaque is defined as a localized thickening >1.2 mm that do not uniformly involve the whole artery. Progression of plaque is defined as an increase in region harboring plaque or number of plaque. Reproducibility of IMT was 0.97. Total plaque area (TPA) will be measured as described before. The plane for measurement of each plaque will be chosen by reviewing the video of the scan to find the largest extent of plaque as seen on the longitudinal view. TPA will be recorded as the sum of the areas of all plaques in the right and left carotid arteries. Reading of the ultrasound scans obtained at baseline and follow-up will be performed concurrently by a single reader (ITC) who is aware of the temporal order of the images but is blinded to all clinical data. The change in TPA will be calculated by subtracting the baseline TPA from the follow-up TPA. The intraobserver intraclass correlation coefficient for TPA was 0.94.

Coronary atherosclerosis assessment CCTA scans will be performed at baseline and 12 months 256-rows multidetector CT (General Electric (GE) Revolution CT) in accordance with the protocol employed in the ACCURACY trial, and will be analysed by an experienced radiologist blinded to clinical data (PT). Coronary artery calcium score (CAC) will be quantified by the Agatston method. The presence, site, stenosis level of plaques will be recorded. Coronary arteries will be standardised to American Heart Association 15-segment model. Segment involvement score (SIS) represented the total number of segments harbouring plaque. Lesions rendering over 50% stenosis of the lumen will be considered as obstructive. For multiple plaques, the most stenotic one will be recorded. Voxels with attenuation less than 130 HU will be assigned to the non-calcified volume of the plaque. For each segment, the presence or absence of 4 coronary artery high risk plaque features will be assessed: positive remodeling, low attenuation plaque, spotty calcification, and the "napkin ring" sign. Positive remodeling is defined as an outer vessel diameter that is 10% greater than the mean of the diameter of the segments immediately proximal and distal to the plaque. Low-attenuation plaque is defined as a focal central area of plaque with an attenuation density of <30 HU. Spotty calcification is defined as focal calcification within the coronary artery wall <3 mm in maximum diameter. The "napkin ring" sign is defined as a central area of low attenuation plaque that had a peripheral rim of high attenuation. Observer agreement for the assessment of coronary artery plaque characteristics has overall been shown to be fair. Plaque volume will be measured automatically based on attenuation (CardIQ Xpress 2.0 Reveal, General Electic).

Toxicity monitoring To monitor the possible side effect of the statin and DMARDs, complete blood count, CK, liver and renal function tests will be performed every visit. Chest X-rays will be obtained at baseline and at the end of the study. The treating physician record all adverse events and serious adverse events and, if necessary, make treatment adjustments in accordance with the protocol. Serious adverse events are defined as any adverse reaction resulting in any of the following outcomes: a life-threatening condition or death, a significant or permanent disability, a malignancy, hospitalization or prolongation of hospitalization, a congenital abnormality, or a birth defect.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilled the Classification of Psoriatic Arthritis (CASPAR) criteria
2. With asymptomatic carotid plaques with <50% stenosis

Exclusion Criteria:

1. History of overt CVD (including myocardial infarction, angina, stroke, and transient ischemic attack)
2. Currently on antiplatelet agents (including aspirin, Clopidogrel etc), or HMG-CoA reductase inhibitors (statins);
3. FRS > 10% at screening visit who are indicated to start statins;
4. had contraindication for statin medication (hypersensitivity to statins, liver disease with transaminase levels of ≥ 2 times the upper limit of normal [ULN], previous statin-induced myopathy or severe hypersensitivity, reactions to other statins
5. Female of childbearing potential who are unwilling to use adequate contraception
6. Pregnant or breastfeeding women
7. Cyclosporine treatment
8. Treatment with medicinal products that have a known interaction with rosuvastatin
9. Uncontrolled hypothyroidism defined as thyroid-stimulating hormone level of >1.5 times the ULN at the first visit [due to the connection between myopathy and hypothyroidism with statin treatment]
10. Secondary hyperlipidemia (primary hypothyroidism, nephrotic syndrome, creatinine level of > 120µmol/l], uncontrolled diabetes mellitus [DM] [glycated hemoglobin >10%], or plasma triglyceride level of >6.8 mmoles/liter [602.3 mg/dl])
11. Other diseases or treatment that reduces the safety of rosuvastatin or treatment that would interfere with use of rosuvastatin (gastrointestinal disease/treatment that may cause malabsorption of rosuvastatin, cancer, severe psychiatric disease, life-threatening ventricular arrhythmias, other medication that increases the risk of rhabdomyolysis, known alcohol abuse, or participation in other studies).
12. Currently on glucocorticoids at a dose >10mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change in CIMT over a period of 12 months between two groups | 12 months
  The change in carotid IMT will be compared between 2 groups. A higher increment indicate greater progression of atherosclerosis

SECONDARY OUTCOMES:
Progression of carotid plaque at 12 months between the two groups. | 12 months
  Progression of carotid plaque at 12 months between the two groups will be analyzed. Plaque progression is an indicator of worsening of carotid atherosclerosis.
Percent change in indexed volume of noncalcified coronary plaque by CCTA over a period of 12 months between the two groups. | 12 months
  Percent change in indexed volume of noncalcified coronary plaque detected by CCTA indicate the coronary atherosclerosis condition in the patient.
Percent change in indexed volume of the sum of fatty plaque and fibrous plaque detected by CCTA over a period of 12 months between the two groups. | 12 months
  Percent change in indexed volume of the sum of fatty and fibrous plaque detected by CCTA indicate the coronary atherosclerosis condition in the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No